CLINICAL TRIAL: NCT01508507
Title: Effectiveness of a Bivalent, Killed Whole-cell Based Oral Cholera Vaccine(Shanchol®) Delivered Through Community-based Mass Vaccination Campaign in a High-risk Population in India: Matched Case-control Studies
Brief Title: Effectiveness of a Bivalent Killed Whole Cell Based Oral Cholera Vaccine
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: International Vaccine Institute (Other)
Collaborators: Department of Health and Family Welfare, Orissa (Other); Regional Medical Research Center, Orissa (Unknown)
Responsible Party: Sponsor
Other Study IDs: CR-WC-10
Record Dates: First submitted 2011-12-14; First posted 2012-01-12 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Cholera
Keywords: Oral; Cholera; Vaccine; Herd; Risk; population; Matched; Control; Case; Bias
MeSH Terms: conditions — Cholera

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Rectal swabs will be collected from all cases that fulfills inclusion criteria. It will be plated directly into TCBS agar as well as after enrichment in APW for 6 to 20 hours (pH 8.6, 37 degree centrigrade). After this overnight incubation, suspected colonies from TCBS will be tested biochemically and agglutinated with polyvalent, Ogawa and Inaba antisera. Biotyping of O1 isolates will be done with chicken erythrocyte agglunitation tests and determination of polymyxin sensitivity. Non - agglunating strains will be tested with antiserum to V cholarae O139 strain. V cholarae isolates will be tested for susceptibility to the following antimicrobials: tetracycline, erythromycin, furazolidin, trimithprim - sulfame thoxale, ciprofloxacin and norfloxacin.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cholera cases group: "Any diarrheal cases or suspected cholera cases from study area, whose stool specimen collected in study health center and examined in reference laboratory, reveals V. cholerae serotype O1/O139 is defined as cholera case"
- Control group: "A randomly selected age matched individual, who have been living in the study area and did not seek care for diarrheal illness in the study health center since vaccination is defined as control"

SUMMARY:
Various field studies has found that the modified , bivalent, whole cell - based oral cholera vaccine (OCV) to be safe, immunogenic and effective with protective efficacy of 67 % in earlier clinical trials. However, the effectiveness of the vaccine in "real" life situation using the public health system is unknown. It is critical to follow up in the same population, where pilot introduction of OCV was introduced and evaluate vaccine proactive effectiveness at individual as well as at population level. The follow - up and determination of effectiveness of mass OCV vaccination was requested by State Government.

DETAILED DESCRIPTION:
The overall goal of this study is to evaluate the protective effectiveness of one or two doses of modified, bivalent, killed whole cell based OCV, given at least 14 days apart, when delivered through community - based mass vaccination campaign using existing public health infrastructure in a high - risk population in Satyabadi block of Puri district, Orissa, India.

This study has following objectives

Primary objectives:

* To evaluate the individual level protective effectiveness of one or two doses of OCV against culture confirmed cholera episodes, severe enough to seek a formal health care.

Secondary objectives:

* To evaluate population - level effectiveness (herd effects)of OCV delivered through a community based mass vaccination when the vaccine is delivered to more than half of population at risk.
* To determine inverse correlation between vaccine coverage and cholera incidence among diverse geographical clusters.

ELIGIBILITY:
Inclusion criteria for cases of the main case-control study are as follows:

* Giving verbal informed consent/assent, or in the case of minors, a parent or guardian give informed consent to participate in the study
* Living in the study area since the start of the mass vaccination
* Submitted a faecal specimen
* Whose residence could be located
* Whose stool specimens yield V. cholera O1 or O139
* Belonging to study population through census database

Exclusion criteria:

* Not giving verbal informed consent/assent, or in the case of minors, a parent or guardian does not give informed consent to participate in the study
* Not living in the study area since the start of the mass vaccination
* No faecal specimen
* Whose residence could not be located
* Whose stool specimens does not yield V. cholera O1 or O139
* Not belonging to study population through census database

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The same population of Satyabadi block, Puri, Orissa, where Pilot introduction of Oral Cholera Vaccine (OCV) was conducted during May - June, 2011. During this campaign, the OCV vaccine was delivered through community based mass vaccination utilizing public health system.
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2013-03; Primary Completion 2014-02 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Vaccine protective effectiveness at individual level | 11 months
  Matched controls will be selected among the persons of the same age group as that of each case. 1 to 4 ratio will be used in matching cases to controls.Information on all other exposure variables will be collected through questionaire interview for both cases and controls."Protective effectiveness (PE) (%) = [1- the odds of vaccination among cholera confirmed cases relative to the odds of vaccination among matched controls] × 100" is the metric to measure vaccine protective effectiveness at individual level.

SECONDARY OUTCOMES:
Population level effectiveness (herd effect) | 11 months
  Indirect effect: Fraction of household members who are vaccinated in households of unvaccinated cases compared with fraction of household members who are vaccinated in households of unvaccinated controls
  Total effect: Fraction of household members who are vaccinated in households of vaccinated cases compared with the fraction of household members who are vaccinated in households of vaccinated controls.
  Overall effects: Fraction of household members who are vaccinated in household of cases compared with fraction of household members who are vaccinated in control households.
Cohort / GIS study for the measure of herd protection | 11 months
  Geographic unit as a cluster for evaluating vaccine herd protection with the use of cohort analysis, using GIS information from the baseline census. Here, there will be comparison in the incidence of the target outcome (cholera or non-cholera diarrhea) according to the level of vaccine coverage of the geographic unit.

CONTACTS AND LOCATIONS:
Overall Officials: Shantanu K Kar, MD, Principal Investigator — Director, Regional Medical Research Center, Bhubanewar, Orissa, India; Thomas F Wierzba, PHD, Principal Investigator — International Vaccine Institute
Locations (1):
- Regional Medical Research Center, Chandrashekharpur, Bhubaneswar, Odisha, India

REFERENCES:
- [Background] Mahalanabis D, Lopez AL, Sur D, Deen J, Manna B, Kanungo S, von Seidlein L, Carbis R, Han SH, Shin SH, Attridge S, Rao R, Holmgren J, Clemens J, Bhattacharya SK. A randomized, placebo-controlled trial of the bivalent killed, whole-cell, oral cholera vaccine in adults and children in a cholera endemic area in Kolkata, India. PLoS One. 2008 Jun 4;3(6):e2323. doi: 10.1371/journal.pone.0002323. PMID 18523643
- [Background] Sur D, Lopez AL, Kanungo S, Paisley A, Manna B, Ali M, Niyogi SK, Park JK, Sarkar B, Puri MK, Kim DR, Deen JL, Holmgren J, Carbis R, Rao R, Nguyen TV, Donner A, Ganguly NK, Nair GB, Bhattacharya SK, Clemens JD. Efficacy and safety of a modified killed-whole-cell oral cholera vaccine in India: an interim analysis of a cluster-randomised, double-blind, placebo-controlled trial. Lancet. 2009 Nov 14;374(9702):1694-702. doi: 10.1016/S0140-6736(09)61297-6. Epub 2009 Oct 8. PMID 19819004
- [Background] Anh DD, Canh DG, Lopez AL, Thiem VD, Long PT, Son NH, Deen J, von Seidlein L, Carbis R, Han SH, Shin SH, Attridge S, Holmgren J, Clemens J. Safety and immunogenicity of a reformulated Vietnamese bivalent killed, whole-cell, oral cholera vaccine in adults. Vaccine. 2007 Jan 22;25(6):1149-55. doi: 10.1016/j.vaccine.2006.09.049. Epub 2006 Sep 29. PMID 17055622
- [Background] Shin S, Desai SN, Sah BK, Clemens JD. Oral vaccines against cholera. Clin Infect Dis. 2011 Jun;52(11):1343-9. doi: 10.1093/cid/cir141. Epub 2011 Apr 14. PMID 21498389